CLINICAL TRIAL: NCT04935294
Title: A Phase I, Open-Label, Parallel Group Study To Evaluate ACH-0144471 Safety, Tolerability, And Pharmacokinetics In Subjects With Normal Renal Function And Subjects With Renal Dysfunction
Brief Title: Study of Danicopan in Participants With Normal Kidney Function and Participants With Kidney Dysfunction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Collaborators: Achillion, a wholly owned subsidiary of Alexion (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ACH471-009
Record Dates: First submitted 2021-06-21; First posted 2021-06-23 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Healthy; Renal Dysfunction
Keywords: Danicopan; ALXN2040; ACH-0144471; Renal Impairment; Pharmacokinetics; Pharmacodynamics; Factor D Inhibitor; Safety
MeSH Terms: conditions — Renal Insufficiency | interventions — danicopan; rhoA GTP-Binding Protein

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: Matched Control Group Of Healthy Participants (Experimental): Participants received a single 200-milligram (mg) treatment on Day 1.
  Interventions: Drug: Danicopan
- Group 2: Severe RI And Not On Dialysis (Experimental): Participants received a single 200-mg treatment on Day 1.
  Interventions: Drug: Danicopan

INTERVENTIONS:
Drug: Danicopan — Oral tablet.
  Other Names: ALXN2040; ACH-0144471 (formerly); ACH-4471; ACH4471; 4471

SUMMARY:
This was an open-label, nonrandomized, multi-center, single-dose, parallel group study to evaluate the effect of severe renal impairment (RI) on the safety, tolerability, pharmacokinetics, and pharmacodynamics of danicopan (ACH-0144471) compared to demographically-matched healthy participants with normal renal function.

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index (BMI) in the range of 18.0 to 40.0 kilograms (kg)/meter squared, inclusive, with a minimum body weight of 50 kg at screening.
* Stable creatinine clearance.

Participants with RI must have met the following additional criteria to be enrolled in this study

* A stable medication regimen was required. Concomitant medications must have been approved by the Sponsor and Investigator (or designee) or pre-specified in the protocol.
* Abnormal laboratory values must not have been clinically relevant at screening or check-in.
* Participants were in good general health at screening and check-in, allowing for the concurrent illnesses associated with chronic kidney disease.
* Stable severe RI.

Healthy matched control participants with normal renal function must have met the following additional criteria to be enrolled in this study

* In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead electrocardiogram, and vital sign measurements at screening or check-in, as determined by the Investigator (or designee).
* Participants had normal renal function.
* Participants must have been demographically matched to a renally impaired participant by age (± 10 years), sex, and BMI (± 20%) at screening.

Key Exclusion Criteria:

* History of any medical or psychiatric condition or disease (aside from RI for RI participants) that might have limited the participant's ability to complete or participate in this clinical study, confound the results of the study, or pose an additional risk to the participant by their participation in the study.
* History of procedures that could alter absorption or excretion of orally administered drugs.
* Body temperature ≥ 38°Celsius on Day - 1 or Day 1 predose; history of febrile illness, or other evidence of infection, within 14 days prior to study drug administration.
* History or presence of drug or alcohol abuse within previous year; current tobacco/nicotine user; positive for alcohol and/or drug screen at screening.
* Participation in any other investigational study drug trial in which receipt of an investigational study drug occurred within 5 half-lives (if known) or 30 days prior to check-in, whichever was longer.
* For matched control participants, use of any prescription medications/products within 14 days prior to check-in and use of any over-the-counter, nonprescription preparations within 7 days prior to check-in, unless deemed acceptable by the Investigator (or designee).
* Donation of whole blood from 3 months prior to study drug administration, or of plasma from 30 days prior to study drug administration; receipt of blood products within 6 months prior to check-in.
* Participant required dialysis within the last 3 months prior to check-in.
* Participant did not produce sufficient urine output to permit urine sampling at screening and/or check-in; history of urinary incontinence prior to check-in.
* History of kidney transplant or actively on a transplant waiting list prior to check-in.
* Any acute or chronic non-renal condition prior to check-in that would have limited the participant's ability to complete or participate in this clinical study.
* Any major surgery within 4 weeks of study drug administration.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2018-05-29 (Actual); Study Completion 2018-05-29 (Actual)

PRIMARY OUTCOMES:
Participants With Treatment-emergent Adverse Events | Day 1 through Day 10 (+/- 2 days)

SECONDARY OUTCOMES:
Area Under The Plasma Concentration-time Curve Extrapolated To Infinity (AUC0-inf) Of Danicopan | Up to 72 hours postdose
Maximum Observed Plasma Concentration (Cmax) Of Danicopan | Up to 72 hours postdose
Time To Reach The Maximum Observed Plasma Concentration (Tmax) Of Danicopan | Up to 72 hours postdose
Alternative Pathway Activity As Measured By Wieslab Assay | Up to 72 hours postdose
Change From Baseline In Plasma Bb Fragment Of Complement Factor B Concentration | Baseline, Up to 72 hours postdose
Change From Baseline In Complement Factor D Concentration | Baseline, Up to 72 hours postdose

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Clinical Trial Site, Miami, Florida
  - Clinical Trial Site, Orlando, Florida
  - Clinical Trial Site, Minneapolis, Minnesota
  - Clinical Trial Site, Saint Paul, Minnesota